CLINICAL TRIAL: NCT06281730
Title: Use of New Generation Fetoscopes in Pregnancies Affected by Fetal Diseases Amenable to Fetoscopy Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mauro H. Schenone, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 23-009197
Record Dates: First submitted 2024-02-21; First posted 2024-02-28 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: In Utero Procedure Affecting Fetus or Newborn
Keywords: Fetoscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Karl Storz fetoscopes (Experimental): Participants will receive In utero surgery using the new generation Karl Storz fetoscopes (11508AAK and 11506AAK) for fetal conditions amenable to treatment with fetoscopy.
  Interventions: Device: Karl Storz New Generation Fetoscope - curved 11508AAK; Device: Karl Storz New Generation Fetoscope - straight 11506AAK

INTERVENTIONS:
Device: Karl Storz New Generation Fetoscope - curved 11508AAK — 11508AAK Miniature straight forward telescope 0-degree set, curved, diameter 3.3 millimeter, length 30 centimeter, 30,000 pixels, autoclavable, irrigation connector, central working channel 4 french, lateral working channel 3 French., remote eyepiece, fiber optic light transmission incorporated.
Device: Karl Storz New Generation Fetoscope - straight 11506AAK — 11506AAK Miniature straight forward telescope 0-degree, straight, diameter 3.3 millimeter, length 30 cm, 30,000 pixels, autoclavable, irrigation connector, central working channel 4 french, lateral working channel 3 french, remote eyepiece, fiber optic light transmission incorporated.

SUMMARY:
The Researchers are trying to determine feasibility and safety of performing surgery in the womb with the Karl Storz fetoscopes (a tool used to access the baby in the body of the mother). This are new and improved fetoscopes that are not yet approved by the FDA.

ELIGIBILITY:
Inclusion Criteria:

* Patient is a pregnant woman 18 and older
* The mother must be healthy enough to have surgery
* The mother must be scheduled for surgery
* Patient provides signed informed consent that details the maternal and fetal risks involved with the procedure

Exclusion Criteria:

* Age <18 years
* Contraindication to abdominal surgery, fetoscopic surgery, or general anesthesia
* Preterm labor, preeclampsia, or uterine anomaly (e.g., large fibroid tumor) in the index pregnancy.
* Fetal aneuploidy, any significant pathogenic or likely significant pathogenic findings on Karyotype or Microarray (if available, but not required), other major fetal anomalies that impacts significantly the fetal/neonatal survival.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-23 (Actual); Primary Completion 2044-02 (Estimated); Study Completion 2044-02 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 12 months
  The count of subjects who experience adverse events
Serious Adverse Events | 12 months
  The count of subjects who experience serious adverse events
Device malfunctions | 12 months
  The number of device malfunction incidents

SECONDARY OUTCOMES:
Mean gestational age at delivery | 12 months
  The mean gestational age at delivery. Measured in weeks.
Successful Completion | 12 months
  The number of successful fetoscopic surgeries in twin twin transfusion syndrome. The measure of success is being able to ablate all anastomoses thought to be involved in causing the twin twin transfusion syndrome.
Satisfaction scores | 12 months
  Surgeon reported satisfaction of the use of the Karl Storz fetoscopes as measured by a 3 item Likert scale questionnaire. The 3 items are scored from 0 - 3, 0 being strongly disagree to 3 being strongly agree. Total scores range from 0 - 9, lower scores indicate less satisfaction, and higher scores indicate more satisfaction.
Live births | 12 months
  The number of subjects to have a live birth following in-utero surgery
Neonatal deaths | 12 months
  The number of subjects who experience a neonate death following in-utero surgery

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Schenone, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No